CLINICAL TRIAL: NCT03920202
Title: Long - Term Bowel Dysfunction Following Low Anterior Resection
Brief Title: Long - Term Low Anterior Resection Syndrome
Acronym: LongLARS
Status: Completed | Type: Observational
Sponsor: National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other)
Responsible Party: Principal Investigator, Audrius Dulskas, Principal investigator, National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos
Other Study IDs: LongLARS
Record Dates: First submitted 2019-02-19; First posted 2019-04-18 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2019-04

CONDITIONS: Bowel; Functional Syndrome
Keywords: Rectal cancer; Bowel dysfunction; Low anterior resection syndrome; Low anterior resection syndrome score; Quality of life
MeSH Terms: conditions — Irritable Bowel Syndrome; Rectal Neoplasms; Intestinal Diseases; Low Anterior Resection Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Data assessing the long-term bowel dysfunction following low anterior resection is still lacking. The aim of this study is to evaluate late functional results of patients who underwent rectal resection for rectal cancer. This included calculating LARS and Wexner score and identifying possible risk factors of late postoperative bowel disorders.

DETAILED DESCRIPTION:
For the last almost 30 years, the gold standard treatment for RC is low anterior resection (LAR) with total mesorectal excision (TME). Unfortunately, up to 80 % of patients undergoing LAR will suffer of bowel dysfunction including faecal urgency, frequent bowel movements, tenesmus or so called Low Anterior Resection Syndrome (LARS). Simply it has been defined as "disordered bowel function after rectal resection, leading to a detriment in quality of life". Same year LARS score was developed. This tool is easy to use and has been internationally and in Lithuania validated. Wexner score is another tool for evaluation of faecal continence.

There are only five studies investigating long-term results after rectal surgery and influence it has on patients' daily life. In one study 47 of 51 patients experienced LARS following ultra-low anterior resection after average 6.5 years. Another study recently reported major LARS in 46% of the patients with the mean median follow-up of 14.6 years. Others showed that 47.5% of patients still experience LARS symptoms at a follow-up period of 13.7 years. Just recently published study assessed bowel function 12 years in patients undergoing rectal resection with or without preventing ileostomy. Authors found that 63 (72%) patients of 87 experienced LARS symptoms with more than a half complaining of major LARS. Moreover, just last year a study published showing that 73% of patients had LARS at first follow up 5 years after the surgery. During the second visit (another 5 years later) same numbers were seen.

The aim of this study was to evaluate late functional results of patients who underwent rectal resection for rectal cancer. This included calculating LARS and Wexner score and identifying possible risk factors of late postoperative bowel disorders.

ELIGIBILITY:
Inclusion Criteria:

* patients diagnosed with rectal cancer without metastasis
* signed consent form
* more than 5 years following the surgery

Exclusion Criteria:

* unwilling to participate
* stage IV disease
* change in operative plan - end colostomy formed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: From 2007 through 2012, we identified a study population of 92 patients with biopsy proven, rectal cancer without distant metastasis located up to 15 cm from anal verge and undergoing low anterior resection with partial or total mesorectal excision. Preoperative staging was performed based on a digital rectal examination, chest and abdominal computer tomography scan (CT), pelvic magnetic resonance imaging (MRI) and colonoscopy with a biopsy.
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-01-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Bowel function assessment using Low anterior resection syndrome questionnaire | 5 years
  Bowel function following low anterior resection surgery for rectal cancer will be assessed using Low anterior resection syndrome score (LARS score - simple 5 question questionnaire). LARS score is a tool consisting of five items, which are as follows: incontinence due to flatus (score range from 0 to 7), incontinence due to liquid stools (score range from 0 to 3), frequency of bowel movements (score range from 0 to 5), clustering (score range from 0 to 11) and urgency (score range from 0 to 16). The severity of each item is calculated on a scale ranging from 0 to 42, with a score of 0-20 (no LARS), 21-29 (minor LARS) and 30-42 (major LARS).

SECONDARY OUTCOMES:
Risk factors: age | 5 years
  Risk factors for having worse bowel function following low anterior resection for rectal cancer - age: older patients (>55years) might have worse bowel function
Risk factors: type of surgical procedure | 5 years
  Risk factors for having worse bowel function following low anterior resection for rectal cancer - type of surgery: rectum resection with total mesorectal excision vs partial mesorectal excision will lead to worse functional outcome.
Risk factors: preoperative chemoradiotherapy | 5 years
  Risk factors for having worse bowel function following low anterior resection for rectal cancer - preoperative chemoradiotherapy might lead to worse functional outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Narimantas Samapavicius, Prof., Study Chair — Klaipėda University
Locations (1):
- National Cancer Institute, Vilnius, Lithuania

IPD SHARING:
Plan to Share IPD: No
Only results of the study will be shared

REFERENCES:
- [Derived] Dulskas A, Kavaliauskas P, Pilipavicius L, Jodinskas M, Mikalonis M, Samalavicius NE. Long-term bowel dysfunction following low anterior resection. Sci Rep. 2020 Jul 17;10(1):11882. doi: 10.1038/s41598-020-68900-8. PMID 32681140